CLINICAL TRIAL: NCT04536597
Title: The Effects of Quince Seed Jelly and Breast Milk on Nipple Fissures During Early Postpartum
Brief Title: Quince Seed Jelly and Breast Milk on Nipple Fissures
Acronym: QSJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Gulbahtiyar DEMİREL, Faculty of Health Sciences, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRSIVAS01
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Primiparity; Postpartum
Keywords: breast milk; early postpartum period; nipple fissures; midwifery; quince seed jelly
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quince seed jelly group (Experimental)
  Interventions: Other: Quince seed jelly group
- Breast milk group (Experimental)
  Interventions: Other: Breast milk group
- Control group (Other): Any kind of application that the mothers in the control group did for the nipple fissures were recorded on the 1st, 3rd, 7th and 10th days postpartum, by the researcher
  Interventions: Other: Control group

INTERVENTIONS:
Other: Quince seed jelly group — Quince seed jelly, prepared by the researcher, was given to the mothers belonging to this group. Briefly, 3 g (2-3 pieces) of quince seeds are placed in 100 mL water and heated to boiling for 10 min. The prepared quince kernel was used for 3 days, immediately after cooling.14,15 On the 1st day postpartum, the researcher provided the mothers with practical training at the hospital, regarding the application of quince seed jelly to the nipple and areola and leaving it to dry. This training was repeated on the 3rd, 7th and 10th days, to ensure that the mothers followed it precisely. The training process was completed in 5-10 min, including questions and answers. Every 3-4 days (days 1, 3, 7 and 10), quince seed jelly prepared by the researcher was given to the mothers to continue applying, according to the procedure. The mothers were asked to apply it after every breastfeeding.
  Arms: Quince seed jelly group
Other: Breast milk group — Mothers in this group received practical training, conducted by the researcher on the 1st day postpartum at the hospital, on applying a few drops of their breast milk to the nipples and areola after each breastfeeding and leaving it to dry. This training lasted 5-10 min. Breast milk application of mothers in this group was recorded on the 1st, 3rd, 7th and 10th days, by the researcher.
  Arms: Breast milk group
Other: Control group — Any kind of application that the mothers in the control group did for the nipple fissures were recorded on the 1st, 3rd, 7th and 10th days postpartum, by the researcher
  Arms: Control group

SUMMARY:
Background: In various experimental or clinical studies, it has been reported that the jelly made from the quince seed is effective in healing wounds (attributed to the antioxidants, which increased fibroblast activity and collagen production, facilitated the formation of granulation tissue and increased blood circulation) and has no side effects or contraindications.

Purpose: To evaluates the effects of quince seed jelly and breast milk on nipple fissures.

Methods: Randomised controlled experimental study.

ELIGIBILITY:
Inclusion Criteria:

* primiparity,
* those having no nipple problems and allergy history
* volunteered to participate in the study

Exclusion Criteria:

* nipple problems and allergy history
* multiparity

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 426 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Nipple pains and fissures | between the 1st and 10th days of the postpartum period
  the Breast Care Monitoring Form

IPD SHARING:
Plan to Share IPD: No